CLINICAL TRIAL: NCT05566704
Title: An Assessment of the Safety and Performance of the Modulus® ALIF System in Patients Undergoing Anterior Lumbar Interbody Fusion
Brief Title: Retrospective Modulus ALIF Study
Status: Completed | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.RMA0222
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis; Stenosis
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Modulus ALIF System
  Interventions: Device: Modulus ALIF System

INTERVENTIONS:
Device: Modulus ALIF System — The Modulus ALIF System is designed to address lumbar pathologies utilizing interbody placement through an anterior or anterolateral surgical approach. The Modulus ALIF System is an interfixated interbody system available in various shapes and sizes to suit the individual pathology and anatomical conditions of the patient.

SUMMARY:
The primary objective of this study is to evaluate the safety and performance of the Modulus ALIF System in patients undergoing anterior lumbar interbody fusion (ALIF) as measured by reported complications, radiographic outcomes, and patient-reported outcomes.

DETAILED DESCRIPTION:
Patients considered for this study will have previously undergone surgery for their spinal condition according to the standard of care of the practitioner. All patients at a given site who meet eligibility requirements will be considered for participation in the study. Available progress notes, medical records, patient-reported outcomes, radiographs (plain film and CT scans, if available), and complications will be obtained from the medical records of all enrolled subjects.

The complication profile and overall performance of the Modulus ALIF System will be assessed using the following:

1. Complications attributable to the use of the Modulus ALIF System as noted in surgical summaries, progress notes, and hospital records; and
2. Radiographic outcome (fusion) and description of device status from available plain film radiographs and CT scan(s); and
3. Neurologic status, symptoms, and/or subject self-reported clinical outcomes (e.g., pain and disability), as available

ELIGIBILITY:
Inclusion Criteria:

1. Availability of progress notes and radiographic information preoperatively and a minimum of 6 months following surgery
2. Male or female patients who are ≥18 years of age at the time of surgery
3. Had undergone a regiment of at least six (6) months of nonoperative care treatment prior to being treated with the Modulus ALIF system, except in patients with progressive neurological deficits, neurogenic claudication causing significant disability, or developed cauda equine syndrome
4. Treated with ALIF procedure with the Modulus ALIF System at:

   * One or two adjacent lumbar and/or lumbosacral levels for degenerative disc disease (DDD), degenerative spondylolisthesis, or spinal stenosis, or
   * Any number of lumbar and/or lumbosacral levels for degenerative scoliosis (defined as >10º coronal curve) or sagittal deformity
5. Supplemental fixation cleared by the applicable regulatory body for use in the thoracolumbar spine unless the procedure meets all of the following criteria:

   * 1-2 levels treated for DDD, and
   * 3 or 4 interfixated screws placed, and
   * Implant lordosis is ≤20°

Exclusion Criteria:

1. Patient was a prisoner at the time of Modulus ALIF treatment
2. Patient was participating in another clinical study during treatment that would confound study data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The analysis population will include all subjects who meet the criteria for enrollment, specifically, those subjects who:
  * Satisfied the inclusion and exclusion criteria
  * Previously underwent the surgical procedure as defined in this protocol
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Rates of complications attributable to the use of the Modulus ALIF System | 12 months
Proportion of subjects with apparent radiographic fusion at 6 months or greater postoperative | 12 months

SECONDARY OUTCOMES:
Change in neurologic status, symptoms, and/or subject self-reported clinical outcomes (e.g., pain and disability), as available | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Malone, MS, Study Director — Globus Medical
Locations (5):
- United States (5):
  - Hoag Orthopedics, Orange, California
  - Girard Orthopedic Surgeons, San Diego, California
  - Georgia Spine & Neurosurgery Center, Atlanta, Georgia
  - OrthoCarolina, Charlotte, North Carolina
  - Atlantic Brain and Spine, Wilmington, North Carolina